CLINICAL TRIAL: NCT01762228
Title: Randomized Controled Clinical Study to Evaluate the Efficacy of the Increase of the Sensorial Stimuli as a Therapeutic Strategy for the Treatment of Elderly Patients With Oropharyngeal Dysphagia.
Brief Title: Efficacy of Two Interventions Increasing Sensory Stimulus in Elderly Patients With Oropharyngeal Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, Pere Clavé, MD, PhD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUTUA-12
Record Dates: First submitted 2012-10-10; First posted 2013-01-07 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Dysphagia
Keywords: Oropharyngeal dysphagia; Elderly; Transcutaneous electrical stimulation; TRPV1 agonist
MeSH Terms: conditions — Deglutition Disorders | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcutaneus electrical stimulation (Active Comparator): Sensorial transcutaneous electrical stimulation to the pharynx and larynx will be used 1 hour/day during 5 days/week for 2 weeks.
  Interventions: Device: Transcutaneous electrical stimulation
- TRPV1 agonist (Active Comparator): Sensorial stimulation of TRPV1 receptors into the oropharynx of patients will be used 3 times/day (before meals) during 5 days/week for 2 weeks.
  Interventions: Dietary Supplement: TRPV1 agonist

INTERVENTIONS:
Device: Transcutaneous electrical stimulation — Using a device which gives electrical stimulation, electrodes will be placed transcutaneously in oropharyngeal muscles of patients giving a sensorial stimuli during one hour for 5 days/week during 2 weeks of treatment.
  Arms: Transcutaneus electrical stimulation
Dietary Supplement: TRPV1 agonist — Patient will be given a TRPV1 agonist natural product (which contains capsaicin) before every meal, during one hour for 5 days/week during 2 weeks of treatment.
  Arms: TRPV1 agonist

SUMMARY:
This study will evaluate with videofluoroscopy (radiologic method to study the deglutitive physiology) the effect on the deglutition of two therapeutic treatments with the duration of 2 weeks, based on the increase of the sensorial stimuli in older patients with oropharyngeal dysphagia:

1. Stimulation of Transient Receptor Potential Vanilloid 1 (TRPV1) oropharynx chanels using a natural agonist administrated in the alimentary bolus.
2. Stimulation of the sensorial neurons of the pharynx and larynx using transcutaneous electrical stimuli.

Moreover, with an electroencephalographic study we will assess the effect of both treatments in the cortical neuroplasticity.

DETAILED DESCRIPTION:
This study will evaluate with videofluoroscopy (radiologic method to study the deglutitive physiology) the effect on the deglutition of two therapeutic treatments with the duration of 2 weeks, based on the increase of the sensorial stimuli in older patients with oropharyngeal dysphagia:

1. Stimulation of Transient Receptor Potential Vanilloid 1 (TRPV1) oropharynx chanels using a natural agonist administrated in the alimentary bolus.
2. Stimulation of the sensorial neurons of the pharynx and larynx using transcutaneous electrical stimuli.

The study will last 5 weeks per patient. At the beginning of the study, patients will receive a videofluoroscopic evaluation and an electroencephalography (evoked potentials) to asses dysphagia and cortical activity of deglutition. After that the first day of the third week they will begin the treatment (group a or b) during 2 weeks. Finally in the fifth week an evaluation of dysphagia will be performed the same way as in week 1 to asses the effects of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (≥70 years) with oropharyngeal dysphagia (OD)
* Patients have to fill in and sign the written informed consent.
* Patients without any of the exclusion criteria.

Exclusion Criteria:

* Patients not able to comply with the protocol.
* Patients currently participating or having participated in another clinical trial in the last 4 weeks.
* Patients with active neoplasia.
* Patients with an active infectious process.
* Patients with severe dementia or inability to communicate.
* Patients with pacemakers.
* Patients with implanted electrodes.
* Patients with epilepsy or convulsive disorders.
* Patients with gastroesophageal reflux disease.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal motor response measured by Videofluoroscopy. | Week 1 and 5.

SECONDARY OUTCOMES:
Cortical activation measured by electroencephalography. | It will be assessed at the beginning and at the end of the study (first and fifth week).

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ortega Fernández, MSc, Principal Investigator — Hospital de Mataró; Pere Clavé, MD, PhD, Study Director — Hospital de Mataró; Laia Rofes, MSc, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró. Consorci Sanitari del Mareme., Mataró, Barcelona, Spain

REFERENCES:
- [Background] Rofes L, Arreola V, Romea M, Palomera E, Almirall J, Cabre M, Serra-Prat M, Clave P. Pathophysiology of oropharyngeal dysphagia in the frail elderly. Neurogastroenterol Motil. 2010 Aug;22(8):851-8, e230. doi: 10.1111/j.1365-2982.2010.01521.x. Epub 2010 Jun 7. PMID 20529208
- [Background] Clave P, Arreola V, Romea M, Medina L, Palomera E, Serra-Prat M. Accuracy of the volume-viscosity swallow test for clinical screening of oropharyngeal dysphagia and aspiration. Clin Nutr. 2008 Dec;27(6):806-15. doi: 10.1016/j.clnu.2008.06.011. Epub 2008 Sep 11. PMID 18789561
- [Background] Jean A. Brain stem control of swallowing: neuronal network and cellular mechanisms. Physiol Rev. 2001 Apr;81(2):929-69. doi: 10.1152/physrev.2001.81.2.929. PMID 11274347
- [Background] Ebihara T, Sekizawa K, Nakazawa H, Sasaki H. Capsaicin and swallowing reflex. Lancet. 1993 Feb 13;341(8842):432. doi: 10.1016/0140-6736(93)93023-t. No abstract available. PMID 8094188
- [Background] Ebihara T, Takahashi H, Ebihara S, Okazaki T, Sasaki T, Watando A, Nemoto M, Sasaki H. Capsaicin troche for swallowing dysfunction in older people. J Am Geriatr Soc. 2005 May;53(5):824-8. doi: 10.1111/j.1532-5415.2005.53261.x. PMID 15877558
- [Background] Caterina MJ, Schumacher MA, Tominaga M, Rosen TA, Levine JD, Julius D. The capsaicin receptor: a heat-activated ion channel in the pain pathway. Nature. 1997 Oct 23;389(6653):816-24. doi: 10.1038/39807. PMID 9349813
- [Background] Hamamoto T, Takumida M, Hirakawa K, Tatsukawa T, Ishibashi T. Localization of transient receptor potential vanilloid (TRPV) in the human larynx. Acta Otolaryngol. 2009 May;129(5):560-8. doi: 10.1080/00016480802273108. PMID 18629672
- [Background] Carnaby-Mann GD, Crary MA. Examining the evidence on neuromuscular electrical stimulation for swallowing: a meta-analysis. Arch Otolaryngol Head Neck Surg. 2007 Jun;133(6):564-71. doi: 10.1001/archotol.133.6.564. PMID 17576907
- [Background] Shaw GY, Sechtem PR, Searl J, Keller K, Rawi TA, Dowdy E. Transcutaneous neuromuscular electrical stimulation (VitalStim) curative therapy for severe dysphagia: myth or reality? Ann Otol Rhinol Laryngol. 2007 Jan;116(1):36-44. doi: 10.1177/000348940711600107. PMID 17305276
- [Background] Gallas S, Marie JP, Leroi AM, Verin E. Sensory transcutaneous electrical stimulation improves post-stroke dysphagic patients. Dysphagia. 2010 Dec;25(4):291-7. doi: 10.1007/s00455-009-9259-3. Epub 2009 Oct 24. PMID 19856025
- [Background] Logemann JA. Dysphagia: evaluation and treatment. Folia Phoniatr Logop. 1995;47(3):140-64. doi: 10.1159/000266348. PMID 7640720
- See also: European Society for Swallowing Disorders — http://www.myessd.org/